CLINICAL TRIAL: NCT05165550
Title: A Phase 1, Double-blind, Placebo-controlled Study of Single Ascending Doses of Elsulfavirine to Evaluate the Safety, Tolerability, and Pharmacokinetics of Elsulfavirine and Its Active Metabolite VM-1500A in Healthy Subjects
Brief Title: Study of Single Ascending Doses of Elsulfavirine to Evaluate the Safety, Tolerability, and Pharmacokinetics of Elsulfavirine and Its Active Metabolite VM-1500A in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HIV-VM1500-10
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: HIV-1-infection
Keywords: HIV-1
MeSH Terms: interventions — elsulfavirine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Elsulfavirine 20 mg. Eight (8) subjects (6 active, 2 placebo) per dose level will be enrolled
  Interventions: Drug: Elsulfavirine
- Cohort 2 (Experimental): Elsulfavirine 40 mg. Eight (8) subjects (6 active, 2 placebo) per dose level will be enrolled
  Interventions: Drug: Elsulfavirine
- Cohort 3 (Experimental): Elsulfavirine 80 mg. Eight (8) subjects (6 active, 2 placebo) per dose level will be enrolled
  Interventions: Drug: Elsulfavirine

INTERVENTIONS:
Drug: Elsulfavirine — Elsulfavirine (Elpida®) 20 mg capsules for oral administration
  Other Names: VM-1500

SUMMARY:
To assess the safety and tolerability of Elsulfavirine following administration of single oral ascending doses in HIV-negative, healthy subjects.

DETAILED DESCRIPTION:
This study is a double-blind, placebo-controlled, outpatient study of single oral ascending doses of Elsulfavirine to evaluate the safety, tolerability, and pharmacokinetics of Elsulfavirine and its active metabolite VM-1500A in HIV-negative, healthy subjects. Eight (8) subjects (6 active, 2 placebo) per dose level will be enrolled. Within each of the three cohorts consisting of 8 subjects, 6 subjects each will receive single oral doses of Elsulfavirine at 20 mg, 40 mg, or 80 mg in an escalating manner, and 2 subjects will receive matching placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-55 years;
2. Good general health as determined by medical history, and by results of physical examination, vital signs, ECG, and clinical laboratory tests obtained within 14 days prior to study drug administration;
3. Body weight ≥ 50 kg and a body mass index of 18.5 30 kg/m2, inclusive;
4. A negative alcohol and drug screen tests;
5. Female subjects must be postmenopausal not less than 2 years, surgically sterile, or if of child-bearing potential, must use two reliable forms of contraception from screening to 3 months after the end of dosing; two reliable forms of contraception include use of condom with spermicide by male partner, or diaphragm with spermicide, or condom use by male partner and diaphragm, or condom use by male partner and non-hormonal intrauterine device.
6. Male subjects must use two reliable forms of contraception from screening to 3 months after the end of dosing; two reliable forms of contraception include condom with spermicide, or diaphragm use by female partner with spermicide, or condom and diaphragm use by female partner, or condom and intrauterine device use by female partner.
7. Ability to comprehend the nature of the study and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire study;
8. Willingness to give written consent to participate after reading the consent form, and after having the opportunity to discuss the study with the investigator or his/her delegate.
9. Willingness to comply to all study procedures and assessments as specified by the protocol.

Exclusion Criteria:

1. Subject participation in more than one treatment group;
2. History or presence of any clinically significant organ system disease, such as chronic cardiovascular, bronchopulmonary, neuroendocrine, musculoskeletal, gastrointestinal, hepatic, renal, blood or skin disease, that could interfere with the objectives of the study or the safety of the subject;
3. Any screening laboratory result outside the normal laboratory reference range and as confirmed upon repeated testing;
4. Presence or history of any abnormality or illness, including gastrointestinal surgery, which in the opinion of the Investigator may affect absorption, distribution, metabolism or elimination of the study drug;
5. Systolic blood pressure less than 90 mm Hg or higher than 130 mm Hg; diastolic blood pressure less than 60 mm Hg or higher than 85 mm Hg; pulse rate less than 60 beats per minute or more than 90 beats per minute;
6. 12-lead ECG with any abnormality or QT/QTc interval of > 450 milliseconds (msec) for men or >470 msec for women;
7. Administration of any prescription drug, over-the-counter drug, or herbal, nutritional, dietary, or vitamin supplement within 14 days of study drug administration, including oral contraceptives; interruption of ongoing oral contraceptive or contraceptive implant birth control is not advised solely for the purpose of this clinical trial participation; Note: Female subjects of child-bearing potential on oral contraceptives or contraceptive implant birth control should discuss this matter with their health care provider.
8. Use of the following prescription medications within 5 half-lives of individual agent or within 28 days prior to enrollment, whichever is longer: corticosteroids by any route, other immunosuppressive therapies, drugs that inhibit cytochrome P450 3A4 (CYP3A4; e.g., ritonavir and other drugs of this class for human immunodeficiency virus [HIV] prophylaxis, ketoconazole, itraconazole or similar azole anti-fungal drugs and macrolide antibiotics such as erythromycin) or the use of any medications that could have a significantly impact on organ function (e.g., barbiturates, omeprazole, cimetidine);
9. Hepatitis B (HBsAg), HIV or Hepatitis C Virus antibodies, positive syphilis test;
10. Positive serum pregnancy test (for women of childbearing potential) at screening or positive urine pregnancy test at Day 1;
11. Acute infections within 4 weeks prior to the screening;
12. Unstable sleep pattern (for instance, night work shifts, sleep disorders, insomnia, recent return from a different time zone, etc.);
13. History of alcohol or drug abuse; alcohol or narcotic consumption within 4 days before the screening and throughout the study, smoking 3 months prior to the screening and throughout the study;
14. Positive allergic anamnesis (including drug intolerance and food allergy), including sensitivity to components of the study medication; Specifically, allergies to sulfa drugs and intolerance to lactose will be exclusionary.
15. Blood/plasma donations (≥450 mL of blood/plasma) within 2 months prior to the screening;
16. Participation in other clinical studies or administration of investigational drugs within 3 months prior to the screening;
17. Any other concurrent medical or major psychiatric condition that makes the subject unsuitable for the clinical study;
18. Employee of the investigational site or the sponsor, who is directly involved in the study, or a family member of such a person.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
The incidence of AEs and SAEs. | 35 days

SECONDARY OUTCOMES:
VM-1500A plasma concentration | 35 days
  Active metabolite plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Brett Smith, MD, PhD, Principal Investigator — Altasciences Clinical Los Angeles, Inc.
Locations (1):
- Altasciences Clinical Los Angeles, Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No